CLINICAL TRIAL: NCT02290665
Title: Localized Therapeutics for the Treatment of Gastrointestinal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sidhartha R Sinha, Principle Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB-29620
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Healthy Adults
Keywords: enema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Thermosensitive gel formulation (Experimental): Thermosensitive gel rectal formulation or saline (control) enema with crossover to the other.
  Interventions: Other: Thermosensitive gel rectal formulation; Other: Saline enema
- Saline enema (Experimental): Thermosensitive gel rectal formulation or saline (control) enema with crossover to the other.
  Interventions: Other: Thermosensitive gel rectal formulation; Other: Saline enema

INTERVENTIONS:
Other: Thermosensitive gel rectal formulation
Other: Saline enema

SUMMARY:
The purpose of this study is to determine the patient preference for a biocompatible thermosensitive solution-gel versus water or saline (liquid) enema. The thermosensitive solution-gel is comprised of poloxamer, an inactive compound that is designated as GRAS (generally recognized as safe) by FDA. It could subsequently be used as a medium for drug delivery. The poloxamer (gel) is administered to study participants in order to assess preference and proximal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Age 18 to 70 years old
* Non-pregnant

Exclusion Criteria:

* GI complaints
* Pregnancy
* Patients with previous colonic surgery or current bowel injury or obstruction
* Allergies to contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2015-09-28 (Actual)

PRIMARY OUTCOMES:
Patient preference, as assessed by questionnaire | Up to 3 hours post-administration

CONTACTS AND LOCATIONS:
Overall Officials: Sidhartha Sinha, MD, Principal Investigator — Stanford University; Aida Habtezion, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States